CLINICAL TRIAL: NCT04540016
Title: A Clinical Trial on Absorption, Metabolism, and Excretion of [14C]HSK7653 in Healthy Adult Male Chinese Subjects - Mass Balance and Biotransformation of [14C]HSK7653 in Human
Brief Title: Mass Balance and Biotransformation of [14C]HSK7653 in Human
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Haisco Pharmaceutical Group Co., Ltd (Industry)
Collaborators: First Affiliated Hospital of Suzhou Medical College (Other)
Responsible Party: Sponsor
Organization: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSK7653-103
Record Dates: First submitted 2020-08-25; First posted 2020-09-07 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Type II Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: A single-center, single-dose, non-randomized, open-label design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm Ⅰ (Other): 25 mg of 80 µCi [14C]HSK7653.
  Interventions: Drug: [14C]HSK7653

INTERVENTIONS:
Drug: [14C]HSK7653 — 25 mg of [14C]HSK7653 (radioactivity of 80 µCi) capsules are taken under fasted condition.

SUMMARY:
A single-center, single-dose, non-randomized, open-label design.

DETAILED DESCRIPTION:
Six healthy adult male subjects will be enrolled and the trial will be carried out in two steps:

Step 1: Two eligible male subjects are enrolled and admitted to the clinical study site after passing verification against inclusion and exclusion criteria on Day -2. After being admitted, the subjects are trained regarding drug administration and urine and stool collection procedures to ensure that they are able to perform relevant operations according to the protocol and SOP requirements. Subjects are deprived of food for at least 10 h and of water for 1 h before drug administration. After oral administration of investigational product in the morning of Day 1 under fasted condition, each subject will be deprived of food for 4 h and of water for 1 h.

Dense sampling is scheduled for all urine and stool samples excreted at specified time intervals within 0-336 h post-dose as well as blood samples at specified time points within 0-336 h post-dose. Sample collection and corresponding safety monitoring will be completed in the morning of Day 15 (the specific time will be decided by the investigator and sponsor based on the phased test results, safety results, and the actual situation) before the subjects leave the phase I clinical trial ward. Subjects will return to the ward on Days 19, 26, 33, and 40 to complete biological sample collection and vital sign monitoring according to protocol requirements. Subjects will return to the ward on Day 47 to complete the last biological sample collection (scheduled to be 1176 h after administration) and various withdrawal examinations according to protocol requirements.

The trial employs phased testing to determine whether the dense sampling and sparse sampling time points should be adjusted and whether collection of blood, urine, and stool samples can be prematurely stopped or should be continued for an extended period based on the test results. If biological sampling duration exceeds 1176 h in this study, then sampling will continue at an interval of 7 days until the protocol-specified evaluation criteria for sampling termination is satisfied. Safety monitoring will continue until the date of sampling completion. The test results in step 1 will be used to determine whether the trial procedure needs to be adjusted.

Step 2: Four eligible male subjects will be enrolled and blood, urine, and stool samples will be collected at specified time points/intervals. The procedures are the same as step 1.

Criteria for sampling termination:

Excretion: The radioactivity of biological samples (urine + stool) collected over two consecutive time intervals from the subject is less than 1% of the dose.

Radioactive blood samples: Plasma radioactivity concentrations at two consecutive time points are < 3 times background plasma concentration.

The target total radioactivity of biological samples (urine + stool) collected from each subject is not lower than 80% of the dose. The investigator should finally determine whether to stop sampling of a subject based on the comprehensive evaluation of radioactive test results, safety results and the actual situation.

The entire trial is based on the complete test samples and data collected from 6 subjects. All subjects must complete the trial procedures according to the protocol requirements during admission in the clinical study site and they are not allowed to leave the clinical study site without permission by the investigator.

Subject may withdraw from the study upon confirmation by the investigator provided that no clinically significant abnormality is observed in clinical observation after completion of the trial. Should any clinically significant abnormality be found, the subject will continue to stay at the study site for observation or leave the study site after comprehensive assessment by the investigator and periodically (usually 7 days from the last test) return to the hospital for retests and followed up until recovery to normal, the abnormality is not clinically significant, or a level deemed acceptable by the investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Chinese males, aged 18-45 years old (inclusive);
2. Body weight ≥ 50.0 kg and body mass index (BMI) between 19.0-26.0 kg/m2 (inclusive);
3. Subjects who voluntarily sign the informed consent form (ICF), able to communicate with the investigator and to complete all trial procedures as per the protocol.-

Exclusion Criteria:

Those who meet any of the following should not be enrolled:

Clinical examination:

1. Clinically significant abnormal results for comprehensive physical examination, vital signs, routine laboratory tests [blood routine, blood biochemistry, coagulation routine, urine routine, stool routine + occult blood, thyroid function, oral glucose tolerance test (fasting blood glucose, 2-hour blood glucose), glycated hemoglobin], visual acuity and ophthalmic examination (slit lamp, introcular pressure, and fundoscopy), 12-lead electrocardiogram (ECG), chest X-ray (anteriorposterior), and abdominal B-ultrasound (liver, gallbladder, pancreas, spleen, and kidney);
2. Positive for hepatitis B surface antigen or E antigen, hepatitis C antibody, HIV antibody, or Treponema pallidum antibodies;

   Medication history:
3. Use of any Western medicine or Chinese patent medicine (including prescription drug, over-the-counter drug, health care product, or live attenuated influenza vaccine) within 14 days prior to screening;
4. Participation in any clinical trial and interference with other investigational drug or medical device within 3 month prior to screening;

   Medical history and surgical history:
5. History of serious clinical diseases or diseases/conditions that the investigator believes may affect the study results, including but not limited to the history of diseases in the motor system, nervous system, endocrine system, circulatory system, respiratory system, digestive system, urinary system, and reproductive system;
6. Past history of organic heart disease, heart failure, myocardial infarction, angina, unexplained arrhythmia, torsades de pointes, ventricular tachycardia, long QT syndrome or symptoms and familial history of long QT syndrome (indicated by genetic evidence or sudden death of a close relative at a young age due to cardiac causes);
7. Have undergone major surgery within 6 months prior to screening or with incomplete healing of the surgical incision; major surgery includes, but is not limited to, any surgery with significant risk of bleeding, prolonged general anesthesia, or incisional biopsy or obvious traumatic injury (excluding cured appendicitis surgery or rectal prolapse surgery);
8. Severe allergic constitution, including known allergy to DPP-4 inhibitors or any excipient of this investigational product (mannitol, microcrystalline cellulose), two or more drugs and food components, or with special dietary requirements and thus unable to follow a standardized diet;
9. With commitment acute/chronic bronchospasm (asthma, chronic obstructive pulmonary disease), pulmonary fibrosis, pulmonary tuberculosis, untreated pneumonitis, or other diseases that affect respiratory function;
10. History of severe hypoglycemic seizure (such as hypoglycemia-induced somnolence, disturbance of consciousness, disorganized speech, or even coma), or history of severe hypoglycemia unawareness;
11. Volunteers judged by the investigator to be unsuitable for participating in this trial for any reason.-

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy Chinese males, aged 18-45 years old (inclusive);
Enrollment: 6 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2021-01-14 (Actual); Study Completion 2021-01-21 (Actual)

PRIMARY OUTCOMES:
Percentage of cumulative drug excretion of [14C]HSK7653 on biological specimens(urine and faeces) accounting for total radiation drug dose | From the start of administration to 50 day after administration
  Though collecting different periods of biological specimens(urine and faeces) , detecting their respective drug excretion of [14C]HSK7653，calculating the total cumulative excretion amount and relevant proportion of each kind of specimen(urine or faeces).
Peak concentration (Cmax) | From the start of administration to 50 day after administration
  Pharmacokinetic Measures
Area under the concentration-time curve (AUC0-t, AUC0-∞) | From the start of administration to 50 day after administration
  Pharmacokinetic Measures

CONTACTS AND LOCATIONS:
Overall Officials: Liyan Miao, PhD, Principal Investigator — Medical Ethics Committee of the First Affiliated Hospital of soochow University
Locations (1):
- the First Affilicated Hospital of Soochow University, Suzhou, China

IPD SHARING:
Plan to Share IPD: No